CLINICAL TRIAL: NCT04578158
Title: A Prospective, Randomized, Open-labelled, Controlled Trial to Study the Adjuvant Benefits of Quercetin Phytosome in Patients With Diagnosis of COVID-19.
Brief Title: Trial to Study the Adjuvant Benefits of Quercetin Phytosome in Patients With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ikram Din Ujjan, MBBS, PhD, Principal Investigator, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUMHS/REC/894
Record Dates: First submitted 2020-10-06; First posted 2020-10-08 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
Keywords: COVID-19, Quercetin Phytosome, Anti-inflammatory, Immunomodulatory, Respiratory distress
MeSH Terms: conditions — COVID-19; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): This arm will receive the standard COVID-19 care as per the hospital physician guidelines.
  Interventions: Drug: Standard COVID-19 care
- Quercetin Phytosome (Experimental): This arm will receive standard COVID-19 care + Quercetin Phytosome
  Interventions: Drug: Standard COVID-19 care; Dietary Supplement: Quercetin Phytosome

INTERVENTIONS:
Drug: Standard COVID-19 care — Patients will receive standard covid-19 care as per the hospital/physician guidelines
Dietary Supplement: Quercetin Phytosome — Patients will receive a daily dose of 400 mg of oral Quercetin Phytosome
  Arms: Quercetin Phytosome

SUMMARY:
The purpose of this study is to investigate if Quercetin Phytosome is beneficial for the treatment of COVID-19.

DETAILED DESCRIPTION:
This is a randomized, open-labelled and controlled study aimed to investigate the adjuvant benefits of Quercetin Phytosome in community-based subjects with confirmed SARS-CoV-2 infection (by RT-PCR). The study has two arms. In one arm the subjects will receive standard COVID-19 care as per the hospital/physician guidelines, whereas in the other arm the subjects will receive standard COVID-19 care + Quercetin Phytosome. The treatment will continue for 30 days. It is proposed that Quercetin Phytosome will contribute to boosting the natural immunity of the subjects and will help in preventing the COVID-19 disease progression i.e preventing the need of hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of either gender
* Confirmed SARS-CoV-2 infection by RT-PCR
* Currently diagnosed with mild-to-moderate symptoms of COVID-19 at home in self-isolation within 3 days of SARS-CoV-2 infection.
* Displaying typical symptoms of COVID-19 such as a high temperature, a new, continuous cough, a loss or change to sense of smell or taste
* Patients who have signed informed consent.

Exclusion Criteria:

* Patients with proven hypersensitivity or allergic reaction to quercetin
* Manifest contrary will

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-03-28 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with COVID-19 disease progression | From day 1 to day 30
  Percentage of subjects who require hospitalisation

CONTACTS AND LOCATIONS:
Locations (1):
- Liaquat University Hospital, Jāmshoro, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Colunga Biancatelli RML, Berrill M, Catravas JD, Marik PE. Quercetin and Vitamin C: An Experimental, Synergistic Therapy for the Prevention and Treatment of SARS-CoV-2 Related Disease (COVID-19). Front Immunol. 2020 Jun 19;11:1451. doi: 10.3389/fimmu.2020.01451. eCollection 2020. PMID 32636851
- [Result] Abian O, Ortega-Alarcon D, Jimenez-Alesanco A, Ceballos-Laita L, Vega S, Reyburn HT, Rizzuti B, Velazquez-Campoy A. Structural stability of SARS-CoV-2 3CLpro and identification of quercetin as an inhibitor by experimental screening. Int J Biol Macromol. 2020 Dec 1;164:1693-1703. doi: 10.1016/j.ijbiomac.2020.07.235. Epub 2020 Aug 1. PMID 32745548
- [Result] Liu X, Raghuvanshi R, Ceylan FD, Bolling BW. Quercetin and Its Metabolites Inhibit Recombinant Human Angiotensin-Converting Enzyme 2 (ACE2) Activity. J Agric Food Chem. 2020 Nov 25;68(47):13982-13989. doi: 10.1021/acs.jafc.0c05064. Epub 2020 Nov 12. PMID 33179911